CLINICAL TRIAL: NCT06350864
Title: High-flow Nasal Cannula (HFNC) Oxygen Therapy Versus Conventional Nasal Oxygen Therapy (COT) in Prolonged Upper Gastrointestinal (UGI) Endoscopy Inside the Intensive Care Unit (ICU): a Prospective, Randomized, Controlled Clinical Study
Brief Title: HFNC Versus Conventional Oxygen Therapy in Prolonged Upper Gastrointestinal Endoscopy in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU R11/2024
Record Dates: First submitted 2024-02-23; First posted 2024-04-05 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-02

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: High-flow Nasal Cannula (HFNC) Oxygen Therapy; Conventional Nasal Oxygen Therapy (COT); Upper Gastrointestinal (UGI) Endoscopy; Intensive Care Unit (ICU); Hypoxia
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hypoxia | interventions — Endoscopy, Digestive System; Endosonography

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, comparative, controlled clinical trial study
Who Masked: Investigator
Masking Description: The patients and anesthesiologists in charge of the case will be unmasked as High-flow nasal cannula HFNC) shape,setting and preparation are completely different from the Conventional nasal oxygen therapy (COT), so masking both of them is impossible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional nasal oxygen therapy (COT) group (35 patients) (Active Comparator): Who will receive 5 L/min oxygen flow through standard nasal cannula (gives FiO2 of about 0.4). The allocated flow rates will be maintained throughout the procedure unless intervention will be required at the discretion of the anesthesiologist in charge of the case.
  Interventions: Device: Conventional nasal oxygen therapy (COT); Device: Upper gastrointestinal endoscopy (UGE) including gastroscopy; Device: Upper gastrointestinal endoscopy (UGE) including Endoscopic ultrasound (EUA)
- High-flow nasal cannula (HFNC) group (35 patients) (Active Comparator): Who will receive 30 L/min oxygen flow through VapothermR Precision Flow HFNC. The fraction of inspired Oxygen (FiO2) will be adjusted at 0.4, temperature at 37◦C with 100% humidity.
  Interventions: Device: High-flow nasal cannula (HFNC); Device: Upper gastrointestinal endoscopy (UGE) including gastroscopy; Device: Upper gastrointestinal endoscopy (UGE) including Endoscopic ultrasound (EUA)

INTERVENTIONS:
Device: High-flow nasal cannula (HFNC) — high flow cartridge and adult size nasal cannula: (flow range: 5-40L/minute, oxygen concentration (FiO2): 21-100%, temperature range: 33-39◦ C, humidity minimum of 12mg/liter)
  Other Names: Vapotherm Precision Flow HI-VNI Technology device
  Arms: High-flow nasal cannula (HFNC) group (35 patients)
Device: Conventional nasal oxygen therapy (COT) — Adult size, single use nasal cannula
  Other Names: Ultramed
  Arms: Conventional nasal oxygen therapy (COT) group (35 patients)
Device: Upper gastrointestinal endoscopy (UGE) including gastroscopy — Upper gastrointestinal endoscopy (UGE) will be either diagnostic and/or therapeutic including variceal band ligation, endoscopic hemostasis as injection of bleeding peptic ulcers with adrenaline or bleeders control via either argon plasma coagulation (APC) or heater probe coagulation.
  Other Names: Pentax Medical 90k series gastroscopy with EPK-P High Resolution Video Process with endoscopic ultrasound (EUS).
Device: Upper gastrointestinal endoscopy (UGE) including Endoscopic ultrasound (EUA) — Upper gastrointestinal endoscopy (UGE) will be diagnostic
  Other Names: Pentax Medical 90k series gastroscopy with EPK-P High Resolution Video Process with endoscopic ultrasound (EUS).

SUMMARY:
Conventional supplemental oxygen therapy (COT) during upper gastrointestinal (UGI) endoscopy via nasal catheter is considered the standard practice in maintenance of oxygenation and prevention of hypoxia. However, it is still unclear if this oxygen delivery method is optimal in a prolonged (more than 15 minutes) procedure in patients admitted to the ICU. Because of shortage of data in this concern, this prospective, randomized, controlled clinical trial study will aim to evaluate and compare the efficacy of high-flow nasal cannula (HFNC) oxygen therapy versus COT in patients who will undergo prolonged either diagnostic or therapeutic UGI endoscopy in the intensive care unit (ICU) .

DETAILED DESCRIPTION:
Study will be conducted in the intensive care units (ICU) of Ain Shams University Hospitals, Cairo, Egypt. Consented and enrolled seventy patients will be randomly assigned to one of the following two groups:

* Conventional nasal oxygen therapy (COT) group (35 patients): Who will receive 5 L/min oxygen flow through standard nasal cannula (gives FiO2 of about 0.4). The allocated flow rates will be maintained throughout the procedure unless intervention will be required at the discretion of the anesthesiologist in charge of the case.
* High-flow nasal cannula (HFNC) group (35 patients): Who will receive 30 L/min oxygen flow through Vapotherm Precision Flow HFNC. The fraction of inspired Oxygen (FiO2) will be adjusted at 0.4,temperature at 37◦C with 100% humidity
* Upper Gastrointestinal (UGI) Endoscopic and anesthetic care as following:
* Pre-procedural full medical and anesthetic history, clinical examination and revision of routine investigations and radiological images will be done.
* Standard monitoring via GE monitor will be connected to the patient as electrocardiogram (ECG) for heart rate (beats/min), pulse oximetry for (SpO2 as a percentage) and non invasive blood pressure (NIBP) (mmHg).
* The intravenous access (IV) will be assessed and flow will be assured
* After positioning the patient in the left lateral position, he will receive either HFNC or COT.
* All UGI endoscopic procedures will be performed by an accredited gastroenterologist. Anesthetic care will be provided by an accredited specialist anesthesiologist. After confirming the readiness of the endoscopist, all patients will undergo deep sedation under monitored anesthetic care with the use of initial slow intravenous (IV) propofol 0.5-1mg/kg over 3-5 minutes which will be titrated to the desired clinical response.Intermittent boluses of 10-20 mg will be used as maintenance and will also be titrated to the desired sedation level. Both the endoscopist and anesthesiologist will be instructed to provide the usual care except for the participant's assigned oxygen delivery device and rate.
* Interventions to change the oxygen delivery rate, Fio2 or even intubation with invasive mechanical ventilation in response to hypoxia will be at the discretion of the anesthesiologist in charge.
* UGI diagnostic and therapeutic endoscopy will be performed by PentaxR Medical 90k series gastroscopy. Therapeutic gastroscopy will include variceal band ligation, endoscopic hemostasis as injection of bleeding peptic ulcers with adrenaline or bleeders control via either argon plasma coagulation (APC) or heater probe coagulation.
* Patients will continue their monitored care in the medical ICU till the control of the causes of their ICU admission or their end.
* Demographics and medical conditions will be collected from the medical records and anesthesiologist assessments. Oxygenation, anesthetic and procedure-related (intraprocedural and shortly post- procedural) data will be collected also. The collected data results will be revised, electronically recorded in datasheet, coded, tabulated, analyzed, and processed using the proper computerized statistical package program. Suitable statistical analysis will be done according to the type of data obtained for each parameter with comparison between both groups to identify any significant differences between them

ELIGIBILITY:
Inclusion Criteria:

* Both males and females with age 20-60 years
* American Society of Anesthesiologists (ASA) class I, II or III
* Patients will undergo UGI endoscopic procedure with anticipated procedure time of over 15 minutes because of complexity of the procedure or recurrence, as assessed by the consultant gastroenterologist responsible for the case

Exclusion Criteria:

* Patient refusal or propofol allergy history.
* Suspected difficult airway or Mallampati score more than 3
* Body mass index (BMI) more than 35 kg/m2 (weight will be measured in kilograms and height in meters,then BMI will be measured by equation where: BMI=weight(Kg) / height square (m2))
* Pregnant patients
* Respiratory compromise as patients dependent on supplemental oxygen including respiratory failure or with active chest condition e.g. bronchial asthma or pneumonia
* Cardiovascular compromise including heart failure and shocked patients
* Severe uncontrolled hematemesis with shocked or risk of aspiration.
* Patients deemed as high risk of SRAEs by the anesthesiologist, anticipated requirement or plan for general anesthesia involving airway instrumentation including a laryngeal mask or tracheal intubation.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Any occurrence of at least moderate hypoxemia of any duration measured by pulse oximetry during the procedure. | During the procedure.
  moderate hypoxemia, defined as SpO2 < 90%

SECONDARY OUTCOMES:
The median lowest SpO2 | During the procedure
  Measured by pulse oximetry during the procedure
Any episode of hypoxia occurring less than 1 minute, from 1 to 5 minutes, or more than 5 minutes | During the procedure
  Hypoxemia may be: mild (SpO2 90%-94%), moderate (SpO2 76%-89%), severe (SpO2 ≤ 75%)
Clinically significant hypoxia | During the procedure
  The need to maneuver the upper airway or to change the flow, Fio2 and/or method of oxygen delivery in response to an episode of hypoxia
Sedation related adverse effects (SRAEs) | During the procedure and immediately after the procedure for 6 hours
  They include hypotension, bradycardia, tachycardia, dysrhythmia, seizure, cardiac arrest, nausea or vomiting, recovery agitation, and delayed recovery
Procedure-related adverse events (PRAEs) | During the procedure and immediately after the procedure for 24 hours
  They include :1. Intra-procedural adverse events: The need to pause or stop the procedure because of an episode of hypoxia, gastrointestinal bleeding requiring intervention or perforation.
  2. Post-procedure adverse events as abdominal pain, bloating or bleeding, throat dryness, headache,gastrointestinal bleeding requiring intervention or perforation.
Propofol total used doses in milligrams (mgs) | During the procedure
  Propofol total used doses during sedation

OTHER OUTCOMES:
Endoscopy procedure time | During the procedure
  The duration of time the endoscope entered until exited the oral orifice.
Anesthetic time | During the procedure
  The duration of time during which intravenous sedation with propofol will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mohamed, MD, Principal Investigator — Ain Shames University
Locations (1):
- Ain Shams University-Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The statistics methods and results data will be shared after completing the study

REFERENCES:
- [Derived] Mohamed AM, Selima WZ. HFNC Oxygen Therapy vs COT in Prolonged Upper Gastrointestinal Endoscopy Inside the ICU: A Prospective, Randomized, Controlled Clinical Study. Indian J Crit Care Med. 2025 Mar;29(3):223-229. doi: 10.5005/jp-journals-10071-24919. Epub 2025 Feb 28. PMID 40110237